CLINICAL TRIAL: NCT00147745
Title: Effects of Colesevelam on Insulin Sensitivity in Type 2 Diabetes Mellitus
Brief Title: Effects of Colesevelam on How the Body Responds to Insulin in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WEL-201
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Results first posted 2009-12-04 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-03

CONDITIONS: Type 2 Diabetes
Keywords: Mechanism of action insulin sensitivity
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Colesevelam Hydrochloride; Insulin Glargine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): colesevelam 3.8g administered daily for 12 weeks
  Interventions: Drug: Colesevelam
- 2 (Placebo Comparator): Colesevelam matching placebo for 12 weeks
  Interventions: Drug: Colesevelam matching placebo
- 3 (Active Comparator): open-label Insulin Glargine for 12 weeks
  Interventions: Drug: Insulin glargine (Lantus)

INTERVENTIONS:
Drug: Colesevelam — Colesevelam 3.8g for 12 weeks
  Arms: 1
Drug: Colesevelam matching placebo — Colesevelam matching placebo for 12 weeks
  Arms: 2
Drug: Insulin glargine (Lantus) — Insulin glargine for 12 weeks
  Arms: 3

SUMMARY:
This study is designed to assess the potential mechanism of action by which WelChol® (colesevelam) may improve blood glucose control in patients with type 2 diabetes

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18 - 75, inclusive
* Diagnosed with type 2 diabetes
* Hemoglobin A1c value greater than or equal to 8.0%
* Antidiabetic treatments may include sulfonylurea agents (non-sulfonylurea agents must be withdrawn)
* Overweight, obese (body mass index 25-45 kg/m2)

Exclusion Criteria:

* Change of dose of lipid or blood pressure lowering therapy within past three months
* Previous treatment with colesevelam for hyperlipidemia
* Serum triglyceride greater than 500 mg/dL
* Serum low density lipoprotein-cholesterol less than 60 mg/dL

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2005-06; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- San Diego VMC, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 21 June 2005 to 22 January 2008 at 3 clinical research sites in the United States of America.
Pre-assignment Details: Subjects were taken off any non-sulfonylurea oral anti-diabetic agents for a period of time appropriate to the drug. Qualified subjects were randomized to colesevelam hydrochloride, placebo, or open-label insulin glargine for 12 weeks. Difficulties enrolling into the insulin group caused the size of this group to decrease from 15 to 6 subjects.
Groups:
- Colesevelam 3.8g: colesevelam 3.8g administered daily for 12 weeks
- Open-label Insulin Glargine: open-label Insulin Glargine for 12 weeks
Period: Overall Study
Arm/Group | Colesevelam 3.8g | Colesevelam Matching Placebo | Open-label Insulin Glargine
Started | 16 | 14 | 6
Completed | 15 | 14 | 6
Not Completed | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Colesevelam 3.8g | Colesevelam Matching Placebo | Open-label Insulin Glargine | Total
Number analyzed (Participants) | 16 | 14 | 6 | 36
Age, Continuous [Mean (Full Range); unit: years] | 55.7 [30 to 71] | 54.0 [38 to 66] | 52.8 [34 to 71] | 54.6 [30 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 1 | 11
  Male | 12 | 8 | 5 | 25
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic | 1 | 2 | 2 | 5
  Black or African American | 5 | 3 | 1 | 9
  White | 8 | 9 | 3 | 20
  Unknown or Not Reported | 2 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 16 | 14 | 6 | 36
Body Mass [Mean (Full Range); unit: kg/m2] | 33.7 [24.6 to 46.1] | 33.7 [27.7 to 44.8] | 35.2 [29.9 to 46.7] | 34.0 [24.6 to 46.7]
Fasting Plasma Glucose [Mean (Full Range); unit: mg/dL] | 162.6 [81 to 208] | 207.9 [135 to 418] | 199.0 [129 to 314] | 186.3 [81 to 418]
HbA1c [Mean (Full Range); unit: percent] | 8.2 [7.1 to 9.8] | 8.5 [7.3 to 10.0] | 9.3 [8.2 to 10.9] | 8.5 [7.1 to 10.9]
Height [Mean (Full Range); unit: cm] | 171.7 [159 to 190] | 168.6 [162 to 187] | 170.8 [157 to 179] | 170.4 [157 to 190]
Weight [Mean (Full Range); unit: kg] | 98.6 [73.2 to 128.5] | 95.8 [72.8 to 130.5] | 103.4 [75.8 to 144.8] | 98.3 [72.8 to 144.8]

OUTCOME MEASURES:

1. Primary Outcome: Difference in Endogenous (Hepatic) Glucose Output During a High-dose Insulin Infusion From Baseline to After 12 Weeks of Treatment.
Description: The parameter measured is the endogenous (hepatic) glucose output during a high-dose insulin infusion. A decrease after treatment with colesevelam is indicative of greater sensitivity of the liver to insulin.
Time Frame: Baseline to 12 weeks
Population: The population analyzed was all randomized subjects who received medication and had a baseline and at least 1 post-randomization assessment of an efficacy variable. One placebo participant did not have a valid post-randomization insulin clamp study. Therefore, the number included in the placebo group for this analysis was 13.
Measure: Least Squares Mean (Standard Error); unit: mg/kg/min
Arm/Group | Colesevelam 3.8g | Colesevelam Matching Placebo | Open-label Insulin Glargine
Number analyzed (Participants) | 15 | 13 | 6
mg/kg/min | -0.06 (0.048) | -0.011 (0.051) | -0.01 (0.076)
Statistical Analysis 1: Comparison: Colesevelam 3.8g vs Colesevelam Matching Placebo; Test type: Superiority or Other; p = 0.5499, ANCOVA; Mean Difference (Final Values) = 0.04, 95% CI [-0.10 to 0.19], Standard Error of Mean 0.070
Statistical Analysis 2: Comparison: Colesevelam 3.8g vs Open-label Insulin Glargine; Test type: Superiority or Other; p = 0.5723, ANCOVA; Mean Difference (Final Values) = -0.05, 95% CI [-0.23 to 0.13], Standard Error of Mean 0.090
Statistical Analysis 3: Comparison: Colesevelam Matching Placebo vs Open-label Insulin Glargine; Test type: Superiority or Other; p = 0.3138, ANCOVA; Mean Difference (Final Values) = 0.09, 95% CI [-0.09 to 0.28], Standard Error of Mean 0.091

2. Primary Outcome: Difference in Endogenous (Hepatic) Glucose Output During a Low-dose Insulin Infusion From Baseline to Week 12.
Description: The parameter measured is the endogenous (hepatic) glucose output during a low-dose insulin infusion. A decrease is indicative of greater senstitivity of the liver to insulin.
Time Frame: Baseline to 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/kg/min
Arm/Group | Colesevelam 3.8g | Colesevelam Matching Placebo | Open-label Insulin Glargine
Number analyzed (Participants) | 15 | 13 | 6
mg/kg/min | -0.08 (0.044) | -0.16 (0.048) | -0.04 (0.070)
Statistical Analysis 1: Comparison: Colesevelam 3.8g vs Colesevelam Matching Placebo; Test type: Superiority or Other; p = 0.2042, ANCOVA; Mean Difference (Final Values) = 0.08, 95% CI [-0.05 to 0.22], Standard Error of Mean 0.065
Statistical Analysis 2: Comparison: Colesevelam 3.8g vs Open-label Insulin Glargine; Test type: Superiority or Other; p = 0.6855, ANCOVA; Mean Difference (Final Values) = -0.03, 95% CI [-0.20 to 0.14], Standard Error of Mean 0.083
Statistical Analysis 3: Comparison: Colesevelam Matching Placebo vs Open-label Insulin Glargine; Test type: Superiority or Other; p = 0.1727, ANCOVA; Mean Difference (Final Values) = 0.12, 95% CI [-0.05 to 0.29], Standard Error of Mean 0.085

3. Secondary Outcome: The Acute Effect of Colesevelam (Multiple Doses) on Oral Glucose Absorption From Baseline to 12 Weeks
Description: The parameter measured is the change in area under the curve for glucose(AUCg) after an oral glucose tolerance test. A decrease in AUCg indicative of drug effect on glucose absorption.
Time Frame: Baseline to 12 weeks
Population: One participant in the colesevelam 3.8g group discontinued. Therefore, 15 participants were included in this analysis.
Measure: Least Squares Mean (Standard Error); unit: mg*hr/dL
Arm/Group | Colesevelam 3.8g | Colesevelam Matching Placebo | Open-label Insulin Glargine
Number analyzed (Participants) | 15 | 14 | 6
mg*hr/dL | -49.1 (36.75) | -4.7 (36.93) | -59.3 (57.27)
Statistical Analysis 1: Comparison: Colesevelam 3.8g vs Colesevelam Matching Placebo; Test type: Superiority or Other; p = 0.4104, ANCOVA; Mean Difference (Final Values) = -44.4, 95% CI [-152.8 to 64.1], Standard Error of Mean 53.17
Statistical Analysis 2: Comparison: Colesevelam 3.8g vs Open-label Insulin Glargine; Test type: Superiority or Other; p = 0.8857, ANCOVA; Mean Difference (Final Values) = 10.1, 95% CI [-132.6 to 152.9], Standard Error of Mean 69.98
Statistical Analysis 3: Comparison: Colesevelam Matching Placebo vs Open-label Insulin Glargine; Test type: Superiority or Other; p = 0.4226, ANCOVA; Mean Difference (Final Values) = -54.5, 95% CI [-191.3 to 82.3], Standard Error of Mean 67.08

4. Secondary Outcome: Change in Hemoglobin A1C Due to Effect of Colesevelam From Baseline to 12 Weeks
Description: The parameter measured is the percent of hemoglobin A that is glycosylated. A decrease in this parameter is indicative of improved glucose control.
Time Frame: Baseline to 12 weeks
Population: One participant in the colesevelam 3.8g group discontinued. Therefore, 15 participants were included in this analysis.
  The least squares mean is adjusted for baseline values. This corrects for differences in baseline values between treatment groups.
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | Colesevelam 3.8g | Colesevelam Matching Placebo | Open-label Insulin Glargine
Number analyzed (Participants) | 15 | 14 | 6
percent | -0.29 (0.258) | 0.16 (0.260) | -0.81 (0.426)
Statistical Analysis 1: Comparison: Colesevelam 3.8g vs Colesevelam Matching Placebo; Test type: Superiority or Other; p = 0.2286, ANCOVA; Mean Difference (Final Values) = -0.45, 95% CI [-1.20 to 0.30], Standard Error of Mean 0.366
Statistical Analysis 2: Comparison: Colesevelam 3.8g vs Open-label Insulin Glargine; Test type: Superiority or Other; p = 0.3184, ANCOVA; Mean Difference (Final Values) = 0.52, 95% CI [-0.53 to 1.57], Standard Error of Mean 0.515
Statistical Analysis 3: Comparison: Colesevelam Matching Placebo vs Open-label Insulin Glargine; Test type: Superiority or Other; p = 0.0613, ANCOVA; Mean Difference (Final Values) = -0.97, 95% CI [-1.99 to 0.05], Standard Error of Mean 0.500

5. Primary Outcome: Acute Effect of a Single Dose of Colesevelam on Oral Glucose Absorption From Baseline to First Dose
Description: Change in area under the curve for glucose (AUCg) after a glucose tolerance test. A decrease in AUCg is indicative of a drug effect.
Time Frame: Baseline (Day -4) to first dose (Day 1)
Population: The entire study population was included in this analysis
Measure: Mean (Standard Deviation); unit: mg*hr/dL
Arm/Group | Colesevelam 3.8g
Number analyzed (Participants) | 36
mg*hr/dL | -38.4 (105.75)
Statistical Analysis 1: Comparison: Colesevelam 3.8g; Test type: Superiority or Other; p = 0.0362, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 12 week treatment period plus 30 days after the last dose of study medication.
Arm/Group | Colesevelam 3.8g | Colesevelam Matching Placebo | Open-label Insulin Glargine
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/14 | 0/6
Other Adverse Events (participants affected / at risk) | 14/16 | 10/14 | 4/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Colesevelam 3.8g (N=16) | Colesevelam Matching Placebo (N=14) | Open-label Insulin Glargine (N=6)
ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 1 | 0 (0)
Constipation (Gastrointestinal disorders) | 6 | 1 | 0 (0)
Diarrhea NOS (Gastrointestinal disorders) | 1 | 1 | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 | 0 (0)
Gastroesophageal Reflux disease (Gastrointestinal disorders) | 1 | 0 (0) | 0 (0)
Vomiting NOS (Gastrointestinal disorders) | 0 (0) | 1 | 0 (0)
Infusion site pain (General disorders) | 0 (0) | 2 | 0 (0)
Oedema (General disorders) | 1 | 1 | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 1
Ear Infection NOS (Infections and infestations) | 1 | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 | 2 | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1
Tooth Abcess (Infections and infestations) | 1 | 0 (0) | 1
Vaginosis Fungal NOS (Infections and infestations) | 0 (0) | 1 | 0 (0)
Viral Infection NOS (Infections and infestations) | 1 | 0 (0) | 0 (0)
Heat exhaustion (Injury, poisoning and procedural complications) | 1 | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 1 | 0 (0) | 0 (0)
Elecrtocariogram ST Segment Depression (Investigations) | 1 | 0 (0) | 0 (0)
Electrocardiogram T Wave Abnormal (Investigations) | 2 | 0 (0) | 0 (0)
Electrocardiogram T Wave Inversion (Investigations) | 0 (0) | 2 | 0 (0)
Heart Rate Increased (Investigations) | 1 | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 (0) | 0 (0)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 | 1
Headache (Nervous system disorders) | 2 | 5 | 1
Migraine NOS (Nervous system disorders) | 0 (0) | 1 | 0 (0)
Dysmenorrhea (Reproductive system and breast disorders) | 0 (0) | 1 | 0 (0)
Erectile Dysfunction NOS (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 (0) | 0 (0)
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Sinus Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If identified by Daiichi Sankyo, Inc. (DSI), any of DSI's confidential information as defined herein shall be deleted…Nothing in this publication section shall be taken as giving DSI any right of editorial control over any publication prepared by Study Site.